CLINICAL TRIAL: NCT00845039
Title: A Randomized Phase II Clinical Trial Investigating Irinotecan Plus Cetuximab With or Without Anti-Insulin-Like Growth Factor-I Receptor Monoclonal Antibody (IMC-A12) for the Treatment of Patients With Metastatic K-Ras Wild Type Carcinoma of the Colon or Rectum That Has Progressed on Oxaliplatin and Bevacizumab Given as First-Line Therapy
Brief Title: A Study of Irinotecan and Cetuximab With or Without IMC-A12 for Treatment of Participants With Colon or Rectum Cancer Who Got Worse After Their First Treatment With Oxaliplatin and Bevacizumab
Acronym: FC-4
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early 22Feb2010 with only 4 participants due to business reasons.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13928; CP13-0708 (Other: ImClone, LLC); I5A-IE-JAED (Other: Eli Lilly and Company); NSABP FC-4 (Other: The National Surgical Adjuvant Breast and Bowel Project)
Record Dates: First submitted 2009-02-10; First posted 2009-02-16 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Tumors; Antibodies, Monoclonal; Colorectal Neoplasms; Metastatic K-RAS Wild-Type Carcinoma of the Colon or Rectum
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Neoplasms; Colorectal Neoplasms | interventions — Cetuximab; Irinotecan; cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetuximab + Irinotecan (Active Comparator): Participants in Treatment Group 1 will receive intravenous infusions of Cetuximab 500 milligrams per square meter (mg/m²) and Irinotecan 180 mg/m².
  Interventions: Biological: Cetuximab; Drug: Irinotecan
- Cetuximab + IMC-A12 + Irinotecan (Experimental): Participants in Treatment Group 2 will receive intravenous infusions of Cetuximab 500 mg/m², IMC-A12 10 milligrams/kilogram (mg/kg) and Irinotecan 180 mg/m².
  Interventions: Biological: Cetuximab; Drug: Irinotecan; Biological: IMC-A12 (cixutumumab)

INTERVENTIONS:
Biological: Cetuximab — Cetuximab 500 mg/m² every 14 days until disease progression or participant intolerance
  Other Names: Erbitux; LY2939777
Drug: Irinotecan — 180 mg/m² every 14 days until disease progression or participant intolerance
  Other Names: Camptosar
Biological: IMC-A12 (cixutumumab) — IMC-A12 10 mg/kg every 14 days until disease progression or participant intolerance
  Other Names: Cixutumumab; LY3012217
  Arms: Cetuximab + IMC-A12 + Irinotecan

SUMMARY:
The purpose of this study is to determine the value of adding IMC-A12 to irinotecan and cetuximab in participants with metastatic colorectal cancer (CRC).

DETAILED DESCRIPTION:
The purpose of this study is to determine the value of adding IMC-A12 to irinotecan + cetuximab in improving progression-free survival (PFS) at 18 weeks from the date of randomization for participants with metastatic Kirsten Rat Sarcoma (K-RAS) wild-type CRC that has progressed on an oxaliplatin/bevacizumab-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Must consent to be in the study and must have signed and dated Institutional Review Board (IRB)-approved consent forms conforming to federal and institutional guidelines for the pre-entry tumor sample submission for central K-RAS testing and for the study treatment
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Must have metastatic CRC
* The CRC tumor or metastatic tumor must be v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog gene (K-RAS) wild-type as determined by central testing
* Must be documented disease progression during first-line therapy containing both oxaliplatin and bevacizumab
* Most recent treatment regimen must have ended ≥21 days prior to randomization, and clinically significant side effects associated with previous therapy must have resolved to ≤Grade 1 with the exception of neuropathy which must have resolved to ≤Grade 2
* Imaging of the chest, abdomen and pelvis with computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 3 weeks prior to randomization
* Must have measurable disease, defined as at least 1 lesion outside a previous radiation therapy (RT) field that can be accurately measured in at least 1 dimension as ≥20 millimeters (mm) with conventional techniques or as ≥10mm with 5mm cuts using a spiral CT scan
* Evidence of adequate bone marrow function: absolute neutrophil (ANC) ≥1200 cubed millimeters (mm³), hemoglobin ≥9 grams per deciliter (g/dL), platelets ≥100,000 mm³
* Evidence of adequate hepatic function. If no liver metastases: aspartate aminotransferase (AST) ≤2.5 times (x) upper limit of normal (ULN), total bilirubin ≤1.5 x ULN for the lab. In the presence of liver metastases: AST ≤5.0 x ULN, total bilirubin ≤1.5 x ULN for the lab
* Serum creatinine must be ≤1.5 x ULN for the lab
* Must have a fasting blood glucose <126 milligrams/deciliter (mg/dL). Fasting is defined as no caloric intake for at least 8 hours

Exclusion Criteria:

* Life expectancy less than 12 weeks
* Diagnosis of anal or small bowel carcinoma
* Tumor that is considered by the surgeon to be amenable to complete resection
* Previous RT to >25% of bone marrow
* RT to sites of measurable disease chosen as target lesions
* Radiological evidence and/or clinical signs or symptoms of central nervous system (CNS) metastases
* Any of the following conditions and events: uncontrolled hypertension, defined as systolic blood pressure (BP) >150 millimeters of mercury (mmHg) or diastolic BP >100 mmHg with or without antihypertensive medication (participants with hypertension that is well-controlled on medication are eligible); unstable angina within 6 months before randomization; New York Heart Association (NYHA) Class III or IV cardiac disease; myocardial infarction (MI) within 6 months before randomization; symptomatic arrhythmia; CNS cerebrovascular ischemia [transient ischemic attack (TIA) or stroke] within 6 months before randomization
* Other malignancies unless the participant is considered to be disease-free and has completed therapy for the malignancy ≥12 months prior to randomization. Participants with the following cancers are eligible if diagnosed and treated within the past 12 months: carcinoma in situ of the cervix, colon carcinoma in situ, melanoma in situ, and basal cell and squamous cell carcinoma of the skin
* Serious or non-healing wound, skin ulcers, or bone fracture
* Any significant bleeding unless the source of bleeding has been resected
* History of bleeding diathesis or coagulopathy (participants on stable anticoagulant therapy are eligible)
* Any evidence of active infection
* Active inflammatory bowel disease
* Grade 3 or 4 diabetes mellitus as defined by National Cancer Institute's (NCI's) Common Terminology Criteria for Adverse Events (CTCAE) v 3.0 pancreatic endocrine: glucose intolerance (participants with diabetes controlled with diet and/or oral medications are eligible)
* Symptomatic interstitial pneumonitis or definitive evidence of interstitial pneumonitis described on CT scan or chest x-ray in asymptomatic participants
* Any other serious concomitant medical condition that, in the opinion of the investigator, would compromise the safety of the participant or compromise the participant's ability to participate in the study
* Previous hypersensitivity reaction to monoclonal antibodies
* Previous treatment with irinotecan, cetuximab, or any agent specifically targeting insulin-like growth factor (IGF) receptors
* Treatment with an investigational drug within 30 days prior to randomization
* Pregnancy or lactation at the time of participant entry
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the participant from meeting the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - ImClone Investigational Site, Vallejo, California
  - ImClone Investigational Site, Greenville, North Carolina
  - ImClone Investigational Site, Scranton, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab + Irinotecan: 500 milligrams per square meter (mg/m²) of Cetuximab administered by intravenous (IV) infusion then followed by 180 mg/m² of Irinotecan by IV infusion on Day 1 of each 14-day cycle until disease progression or participant intolerance.
- Cetuximab + IMC-A12 + Irinotecan: 500 mg/m² of Cetuximab administered by IV infusion then followed by 10 milligrams per kilogram (mg/kg) of IMC-A12 IV followed by 180 mg/m² of Irinotecan by IV infusion on Day 1 of each 14-day cycle until disease progression or participant intolerance.
Period: Overall Study
Arm/Group | Cetuximab + Irinotecan | Cetuximab + IMC-A12 + Irinotecan
Started | 2 | 2
Received at Least 1 Dose of Study Drug | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Cetuximab + Irinotecan: 500 mg/m² of Cetuximab administered by IV infusion then followed by 180 mg/m² of Irinotecan by IV infusion on Day 1 of each 14-day cycle until disease progression or participant intolerance.
- Cetuximab + IMC-A12 + Irinotecan: 500 mg/m² of Cetuximab administered by IV infusion then followed by 10 mg/kg of IMC-A12 IV followed by 180 mg/m² of Irinotecan by IV infusion on Day 1 of each 14-day cycle until disease progression or participant intolerance.
- Total: Total of all reporting groups
Arm/Group | Cetuximab + Irinotecan | Cetuximab + IMC-A12 + Irinotecan | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 52.0 [48 to 56] | 59.5 [56 to 63] | 55.8 [48 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Rate at 18 Weeks
Time Frame: Approximately 18 Weeks
Population: Zero participants analyzed. Per Clinical Study Report, decision made by ImClone and NSABP at time of study closing to not perform summary analysis on N= 4 due to validity of data related to low number of participants and concerns on maintaining participant confidentiality for low number of participants.
Groups:
- Cetuximab + IMC-A12 + Irinotecan: 500 mg/m² of Cetuximab administered by IV infusion then followed by 10 mg/kg of IMC-A12 IV followed by 180 mg/m² of Irinotecan by IV infusion on Day 1 of each 14-day until disease progression or participant intolerance.
Arm/Group | Cetuximab + Irinotecan | Cetuximab + IMC-A12 + Irinotecan
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Objective Response Rate (ORR) [Complete Response (CR) + Partial Response (PR)]
Time Frame: Randomization up to 26.3 months
Population: as for outcome 1
Arm/Group | Cetuximab + Irinotecan | Cetuximab + IMC-A12 + Irinotecan
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Time Frame: Randomization up to 26.3 months
Population: as for outcome 1
Arm/Group | Cetuximab + Irinotecan | Cetuximab + IMC-A12 + Irinotecan
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression Free Survival (PFS) Over Entire Duration
Time Frame: Randomization up to 26.3 months
Population: as for outcome 1
Arm/Group | Cetuximab + Irinotecan | Cetuximab + IMC-A12 + Irinotecan
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: The Number of Participants Who Had a Complete Resection/Ablation of Metastases With no Evidence of Disease Remaining (Resection Rate)
Time Frame: Randomization up to 26.3 months
Population: as for outcome 1
Arm/Group | Cetuximab + Irinotecan | Cetuximab + IMC-A12 + Irinotecan
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Toxicity of the Irinotecan + Cetuximab + IMC-A12 Regimen
Time Frame: Randomization up to 26.3 months
Population: as for outcome 1
Arm/Group | Cetuximab + IMC-A12 + Irinotecan
Number analyzed (Participants) | 0

7. Secondary Outcome: Post-treatment Serum Levels of IMC-A12 in Participants Receiving IMC-A12
Time Frame: Prior to infusion at Cycles 1, 4, 7 (2-week cycles), and 4 to 6 weeks following discontinuation of treatment IMC-A12 up to 77 weeks
Population: as for outcome 1
Arm/Group | Cetuximab + IMC-A12 + Irinotecan
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Behavioral and Health Outcomes [BAHO] Quality of Life (QoL) Questionnaire
Time Frame: Baseline, after Cycle 3 (14-day cycle), study discontinuation 30-day follow-up (up to 26.3 months)
Population: as for outcome 1
Arm/Group | Cetuximab + Irinotecan | Cetuximab + IMC-A12 + Irinotecan
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Serum Anti-IMC-A12 Antibody Assessment
Time Frame: as for outcome 7
Population: as for outcome 1
Arm/Group | Cetuximab + IMC-A12 + Irinotecan
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: The Number of Participants Who Died During 30-Day Follow-Up
Description: Reported are the deaths during the 30-day follow-up period regardless of causality.
Time Frame: 26.3 months post-randomization up to 30-day post-treatment follow-up
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab + Irinotecan | Cetuximab + IMC-A12 + Irinotecan
Number analyzed (Participants) | 2 | 2
Participants | 1 | 1

ADVERSE EVENTS:
Arm/Group | Cetuximab + Irinotecan | Cetuximab + IMC-A12 + Irinotecan
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab + Irinotecan (N=2) | Cetuximab + IMC-A12 + Irinotecan (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab + Irinotecan (N=2) | Cetuximab + IMC-A12 + Irinotecan (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (4) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (2)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated early 22Feb2010 with only 4 participants due to business reasons. Data were collected for too few participants to draw statistically meaningful conclusions and included concerns on participant confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.